CLINICAL TRIAL: NCT07117617
Title: Effects of Inertial Load of Water on Lower Extremity Joint Moments During Landing and Cutting
Brief Title: Effects of Inertial Load of Water on Lower Limb Joint Moments During Landing and Cutting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ja Yeon Lee (Other)
Responsible Party: Sponsor-Investigator, Ja Yeon Lee, Principal Investigator, Busan University of Foreign Studies
Organization: Busan University of Foreign Studies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUFS-DST-2025
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers; Physical Fitness; Lower Extremity
Keywords: Inertial load of water; Dynamic Stability Training; Joint Moments; Landing and Cutting

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either a control group or an experimental group undergoing water-based perturbation training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inertial load of water Training (Experimental): Participants in this group performed dynamic stability training using a water-filled bag (AquaBag) for 10 weeks to improve lower limb Joint moments during landing and cutting tasks.
  Interventions: Behavioral: Dynamic Stability Training with Inertial load of water
- Control (No Intervention): Participants in this group did not receive any training intervention during the 10-week study period.

INTERVENTIONS:
Behavioral: Dynamic Stability Training with Inertial load of water — A 10-week training program using AquaBag to enhance lower limb joint stability and neuromuscular coordination. Exercises included dynamic stepping, lunging, and landing tasks under water load-induced perturbations.
  Arms: Inertial load of water Training

SUMMARY:
This study examined whether a 10-week dynamic stability training program using water-filled equipment could improve joint control and postural stability during landing and directional changes.

Twenty-six healthy young men were randomly assigned to either a training group, which performed water-based exercises, or a control group, which did not receive any intervention.

All participants performed a landing followed by a 90-degree cutting task, and joint moment data were collected using a 3D motion capture system.

The study aimed to determine if water-based perturbation training enhances neuromuscular control and reduces biomechanical stress during complex movements.

DETAILED DESCRIPTION:
The purpose of this study was to investigate the effects of dynamic stability training using the inertial load of water on lower limb joint moments and postural control during landing and subsequent 90-degree directional changes. Rapid deceleration and cutting movements are known to generate high biomechanical loads on the lower extremities, especially during transitions from the non-dominant to dominant leg. Enhancing neuromuscular control in these situations may help reduce injury risk and improve movement efficiency.

A total of 26 healthy male participants in their 20s were recruited and randomly assigned to either an experimental group (n = 13) or a control group (n = 13). The experimental group completed a 10-week training program using water-filled bags designed to induce dynamic perturbation and promote balance and joint control. The control group did not undergo any training intervention during the same period.

All participants performed a standardized movement task consisting of single-leg landing followed by a 90-degree cutting maneuver. A 3D motion capture system and force plates were used to collect data on joint moments and biomechanical responses during both the landing and change-of-direction phases. Pre- and post-intervention data were compared to determine the effectiveness of the water-based perturbation training.

This study was designed to evaluate whether unstable load training can serve as an effective method for improving lower extremity biomechanics and dynamic stability in young adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males aged 20-29 years
* No history of musculoskeletal injury or surgery in the past 6 months
* No neurological or balance disorders
* Right-leg dominant

Exclusion Criteria:

* Participation in any other structured training program during the study period
* Any current or chronic pain affecting physical activity
* Use of medications that affect balance or neuromuscular control

Ages: 20 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Peak Joint Moment of the Lower Extremity During Landing and Cutting | Baseline and after 10 weeks of intervention
  This outcome includes the peak moments of the hip, knee, and ankle joints in all three planes (sagittal, frontal, and transverse) measured during the landing and subsequent 90-degree change-of-direction task. The values are derived using a 3D motion capture system to calculate inverse dynamics.

CONTACTS AND LOCATIONS:
Overall Officials: Ja Yeon Lee, PhD, Principal Investigator — Department of Sports and Health Convergence
Locations (1):
- Busan University of Foreign Studies, Busan, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared because data sharing was not included in the participants' consent.